CLINICAL TRIAL: NCT00604526
Title: Pilot Study of High Dose Rate Prostate Brachytherapy as Salvage for Locally Recurrent Prostate Cancer Previously Treated With External Beam Radiotherapy
Brief Title: High Dose Rate Prostate Brachytherapy as Salvage for Locally Recurrent Prostate Cancer Previously Treated With External Beam Radiotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-122
Record Dates: First submitted 2008-01-08; First posted 2008-01-30 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Prostate Cancer
Keywords: recurrent
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence

ARMS (1):
- 1 (Experimental): Questionnaires, Iridium 192 radioactive seeds
  Interventions: Radiation: High dose rate (HDR) brachytherapy using Iridium 192 radioactive seeds

INTERVENTIONS:
Radiation: High dose rate (HDR) brachytherapy using Iridium 192 radioactive seeds — Pre-tx Sexual function questionnaire Quality of Life baseline, Treatment with HDR (Two days) Treatment: Iridium 192 radioactive seeds temporarily inserted into patient. Post treatment (after HDR) Month 1 (+/- 2 weeks), 3 (+/- 1 month), 6 (+/- 1 month), 9 (+/-1 month), 12 (+/- 1 month)* NCI CTC GU and GI assessment,IPSS, IIEF, PSA lab test, Prostate HRQOL
  *After 1 year, will follow up with doctor about every 6 months.

SUMMARY:
High dose rate (HDR) brachytherapy is a form of radiation treatment using temporary radioactive seeds. This is done by placing very tiny catheters or tubes into the prostate and then inserting temporary radioactive seeds, called Iridium 192, through these catheters. HDR brachytherapy gives precise radiation to the prostate with less radiation given to the normal tissues near the prostate. For patients who have been treated with external beam radiation to the prostate before, HDR brachytherapy can give radiation again to the prostate without exposing the normal tissues around the prostate to significantly more radiation. This may be safer than giving external beam radiation again. The purpose of this study is to test the safety of high dose rate temporary brachytherapy (HDR) for prostate cancer that has come back after external beam radiation. We want to find out what effects, good and/or bad, the treatment has on you and your recurrent prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* KPS > than or equal to 80
* Able to give informed consent
* Able to complete toxicity scales and questionnaires
* Histologically MSKCC confirmed diagnosis of recurrent prostate cancer.
* Documented history of definitive radiotherapy to the prostate gland
* IPSS of < than or equal to 15 at the time of evaluation
* PSA < than or equal to 15 ng/ml
* Organ confined disease

Exclusion Criteria:

* Unable to tolerate general anesthesia
* Abnormal complete blood count. Any of the following:
* Platelet count less than 75,000/ml
* Hb level less than 10 gm/dl
* WBC less than 3.5/ml
* Abnormal coagulation profile:
* INR > 2.5
* Abnormal Liver function tests (>1.5 x normal value)
* Abnormal renal function tests (creatinine > 1.5)
* Evidence of metastatic disease (bone scan, radiographs, MRI findings)
* Prostate volume > 50 cc
* Unable to meet treatment planning criteria
* History of rectal surgery
* External beam radiation dose to the prostate > 86.4 Gy if standard treatment planning dose constraints were met
* History of inflammatory bowel disease
* Expected survival < 1 year
* Unable to undergo bone scan, CT or MRI evaluation
* Unavailable for regular follow up

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
assess feasibility & toxicity of HDR as salvage ther for local recurrent prostate cancer after ext beam radiotherapy. QOL instruments and questionnaires including the MSK prostate QOL instrument, the IIEF, IPSS , & the NCI CTC is used to assess toxicity. | conclusion of study

SECONDARY OUTCOMES:
To assess biochemical or PSA relapse free survival. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiya Yamada, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org